CLINICAL TRIAL: NCT05397067
Title: Implementation of Low Cost Solutions to Help Facilitate Linkage to Care for Persons with Hepatitis C Virus Infection
Brief Title: Linkage to Care for Persons with Hep C Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Mariana Gomez, Principal Investigator, Carilion Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-21-1472; UL1TR003015 (NIH)
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis C, Chronic; Substance Use Disorders
Keywords: Hepatitis C; Substance use disorder; Linkage to care
MeSH Terms: conditions — Hepatitis C, Chronic; Substance-Related Disorders; Hepatitis C

STUDY DESIGN:
Intervention Model Description: Two types of intervention will be tested. The first is the provision of a Peer Specialist (PS), and the second is the use of vouchers (food, transportation, phone)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer specialist and Vouchers (Experimental): Intervention arm
  Interventions: Behavioral: Peer specialist (PS) and vouchers
- Standard of care (No Intervention)

INTERVENTIONS:
Behavioral: Peer specialist (PS) and vouchers — this participants will receive vouchers from PS
  Arms: Peer specialist and Vouchers

SUMMARY:
Hepatitis C Virus (HCV) infection is an ongoing challenge in the United States, with an estimated 2.4 million individuals living with HCV in 2016. According to the Virginia Department of Health, over 11,500 people were living with HCV infection in 2017 with a rate of 170 reported cases/100,000 adults. This same year, the situation was even more dire in Roanoke City which had a rate of 524/100,000 adults. Treatment with antiviral medication is curative and well tolerated. However, gaps remain in the ability of the health system to engage the most vulnerable patients to start and complete treatment. People with HCV infection usually are unaware of the infection, which allows the disease to progress to liver damage, liver cancer and death if left untreated.At each stage of the screening, testing, and treatment process, there is significant patient loss to follow-up. Drop-off most commonly occurs between diagnosis and the first visit to a treating provider.

Key barriers to successful engagement include: 1) communication issues, such as lack of phone or limited phone access; 2) lack of transportation; 3) significant social issues such as poverty; 4) substance use disorder; and 5) a limited understanding of the consequences of untreated HCV infection. In this mixed-method design, the investigators propose a pilot study that will provide education and resources, such as vouchers for phone, transportation, and meals, to the most vulnerable patients that will facilitate engagement in treatment as additional factors that may influence dropout rates are evaluated.

DETAILED DESCRIPTION:
Aim 1: To identify perceived barriers and facilitating factors to completion of HCV treatment by patients and providers at a local level.

The investigators will conduct a qualitative study, informed by current literature, asking patients with a new diagnosis of HCV infection, patients with a history of HCV infection, and providers who specialize in HCV treatment about their perceptions of barriers and facilitators to treatment.

Aim 2: To pilot simple solutions to known basic social problems affecting communication and access to HCV infection care, leveraging peer counselors who are trained in engaging and retaining patients with HCV infection in treatment by bringing earlier, language-appropriate education to patients, while facilitating the LTC process. The investigators will provide time for a Peer Specialist (PS) and vouchers (e.g., for phones, meals, and transportation) to patients at the point of their initial test. The investigators will specifically target people with substance use disorder (PWSD) as our population for this study.

Aim 3: To identify other system-based interventions to address those barriers and optimize the things that will facilitate care and LTC.

The investigators will conduct a local "call-to-action" to leverage local data on the incidence, prevalence, morbidity, and mortality associated with HCV infection, and the findings of our qualitative analysis from specific Aim 1, to identify actionable, sustainable interventions to increase adherence to HCV infection screening, testing, and treatment through systems improvement.

This project seeks to determine whether the interventions (PS, vouchers) influence individual attendance at the first treatment appointment. In addition, what additional factors might be influencing individuals to adhere to their first appointment. Do these individuals find the interventions useful? What other barriers exist?

The investigators will use a mixed methods approach to address these questions. A mixed methods approach was chosen because the quantitative data will allow the investigators to perform descriptive and inferential statistics. The qualitative data will add a richness to our understanding of why our interventions may or may not prove successful.

Qualitative study: This study will help the investigators to understand the extent to which interventions are adopted and what barriers to adoption might exist. The investigators plan to conduct semi-structured key informant interviews with 10 patients and 10 care providers. Interviews will last approximately 30 minutes. Barriers and facilitators (or perceived barriers and facilitators for care providers) to attendance at the first treatment appointment, will be discussed. It is anticipated to use the social-ecological model as a framework and will use axial coding for analysis. The output of this aim is anticipated to be a list of barriers and facilitators (Aim 1). The output of this aim will help to frame additional intervention studies in the future (Aim 3).

Quantitative study: Two types of intervention will be tested. The first is the provision of a PS, and the second is the use of vouchers (food, transportation, phone) to facilitate LTC. These two interventions are linked in this study (see limitations section). Our hypothesis is that this intervention will lead to a greater likelihood of the individual attending their first treatment appointment. Individuals that have a new diagnosis of HCV infection from the Carilion Clinic system will be provided a PS and specific vouchers based on the specialist's assessment of their specific needs at the time of their initial diagnosis. PS's work from the perspective of their lived experience with mental illness/substance use disorder and recovery. Being a PS requires being open about having been diagnosed with a mental illness or substance use disorder. This openness is to help educate others about the reality and the possibility of recovery. The investigators plan to work with them to help patients with substance use disorders and HCV infection to engage in the benefits of HCV treatment as well as to facilitate LTC.

The investigators will use a pragmatic trial (quasi-experimental) approach; specifically, an interrupted time-series design (3 phases) and analysis. The investigators will compare a sample of individuals newly diagnosed with HCV infection pre-implementation to a post-implementation sample, with a short washout period in the middle (phase 1-pre; phase 2-washout; phase 3-post). This is a between-subjects design. Our main measure of interest is attendance at the initial treatment appointment. Although an accurate power calculation is difficult, it is estimated that for an effect size of 2, an n of 36 per phase (36 pre and 36 post), should allow for detection of a 0.05 significant difference between pre- and post-implementation.19 This calculation is based on an assumption of no auto-correlation. The investigators anticipate using an ANOVA for statistical comparisons. The output of this analysis will be a preliminary test of the relationship of our intervention and attendance at the first treatment appointment. Since this is a pilot proposal, designed to build collaboration and ensure our processes are reliable, the investigators will also gather qualitative data on the process of giving out vouchers, the availability and use of the PS, and any other process variables of interest (Aim 3).

ELIGIBILITY:
Inclusion criteria:

* 18 years or older, positive Hepatitis C antibody test,
* elevated Hepatitis C RNA
* history of substance use disorder

Exclusion criteria:

* under 18 years old,
* history of treatment of Hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Attendance at first appointment | Through study completion, an average of 6 months
  Attendance at first appointment for HCV treatment will be compared between the control and intervention arms

OTHER OUTCOMES:
Semi-structured qualitative interviews | Interviews will be conducted through study completion, an average of 6 months for the selected participants and care providers. Interviews will be collected throughout the study.
  10 participants and 10 care providers undergo interviews to determine additional barriers and facilitators to HCV care. The output of these interviews will be a list of barriers and facilitators to care.

CONTACTS AND LOCATIONS:
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No